CLINICAL TRIAL: NCT02196090
Title: Application of Vagal Stimulation by Cold Face Mask in Exposure and Response Prevention for Obsessive Compulsive Disorder
Brief Title: Application of Vagal Stimulation in Exposure and Response Prevention for Obsessive Compulsive Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SLAM-RD-001
Record Dates: First submitted 2014-06-24; First posted 2014-07-21 (Estimated); Last update posted 2016-02-29 (Estimated); Status verified 2016-02

CONDITIONS: Obsessive Compulsive Disorder
Keywords: OCD, Exposure and Response Prevention, Vagal Stimulation
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single arm (Experimental): Study uses the single case series design with only one arm. All participants in the one arm will have procedures with treatment as usual (Exposure and Response Prevention) alternating with procedures including the vagal maneuver (Cold Face Gel Mask).
  Interventions: Behavioral: Exposure and Response Prevention; Device: Cold face gel mask

INTERVENTIONS:
Behavioral: Exposure and Response Prevention — A procedure where patients with OCD test out their fears without responding by compulsive act.
  Other Names: ERP
Device: Cold face gel mask — Temporary application of cold eye mask on the face is commonly used for relaxation purpose.

SUMMARY:
Obsessive Compulsive Disorder (OCD) is a condition associated with recurrent intrusive distressing thoughts, images and urges compelling the person to perform neutralizing acts or thoughts to the extent of significantly interfering with their daily activities. The symptoms of OCD are associated with both subjective and objective signs of distress. Treatment for Obsessive Compulsive Disorder is often associated with significant subjective distress with high dropout rates and often only limited improvement. Attempts to reduce distress in anxiety often focus on re-establishing the sympathovagal balance by enhancing the vagal or parasympathetic tone and it has been suggested that this can reduce the mobilization behaviours of fight or flight response and improve emotion regulation. This study will investigate the effect of a procedure potentially reducing distress and improving outcome of treatment in inpatients admitted for treatment for OCD to the Anxiety Disorders Residential Unit. The procedure will be based on increasing vagal tone by application of cold face mask on 3 consecutive days in addition to the standard Exposure and Response Prevention therapy (ERP).

DETAILED DESCRIPTION:
1. Background

   Obsessive Compulsive Disorder (OCD) is a condition associated with recurrent intrusive distressing thoughts, images and urges compelling the person to perform neutralizing acts or thoughts to the extent of significantly interfering with their daily activities. The symptoms of OCD are associated with both subjective and objective signs of distress. Psychophysiological studies of OCD and other anxiety disorders often report abnormal sympathovagal balance with decreased parasympathetic or vagal tone and increased sympathetic tone (Hoehn-Saric et al 1995, Broderick et al 2013, Kawano et al 2012, Pittig et al 2013, Buhlmann et al 2007, Blechert et al 2007, Friedman and Thayer 1998).

   The first line treatment of OCD is Cognitive Behaviour Therapy (CBT) which includes Exposure and Response Prevention (ERP) when the patient tests out their fears without responding by compulsive act (NICE Clinical Guideline 31). ERP treatment itself is often associated with significant subjective distress (Kellner et al 2012) with dropout rates up to 20% and only minimal improvement in another 20% of patients (Foa 2010). Various modalities of treatment reducing the subjective and physiological distress have been used in treatment of anxiety disorders and symptoms (Streeter et al 2012, Miu et al 2009, Gorman et al 2000) and similar approach could increase the rates of improvement and adherence to ERP treatment in OCD. Most of the attempts to reduce distress in anxiety focus on re-establishing the sympathovagal balance by enhancing the vagal or parasympathetic tone and it has been suggested that this can reduce the mobilization behaviours of fight or flight response and improve emotion regulation (Austin et al 2007). Disgust is an emotion implicated to have significant role on anxiety disorders such as OCD with contamination fears (Moretz and McKay 2008). It has been shown to have only limited response to exposure therapy (Olatunji et al 2009) and can be associated with increased avoidance and reduced compliance with exposures (Olatunji et al 2007) possibly contributing to poorer treatment outcome. Disgust can be associated with changes in sympathovagal balance (Ottaviani et al 2013) but the effect of manoeuvres affecting this balance has not been tested.

   Vagal tonus can be increased with specific procedures called vagal manoeuvres. These include the diving reflex, Valsalva manoeuvre, pressure on the eyeball and carotid sinus massage, with the diving reflex being one of the most effective (Arnold 1999). The diving reflex is a phylogenetically ancient physiological phenomenon believed to facilitate survival after immersion in cold water through bradycardia and peripheral vasoconstriction redistributing blood flow to vital organs (Gooden 1994). The combined bradycardia and vasoconstriction effect indicates on complex sympathovagal activation and the bradycardia itself is believed to be due to central vagal activation (Stemper et al 2002). The natural trigger for diving reflex includes change in body position, apnoea and sensation of cold and wet surface on the face and a cold sensation on the face is sufficient to induce the vagal response. This is believed to be transmitted by the ophthalmic branch of the trigeminal nerve and can be achieved by using cold compressions or cold face gel masks (Khurana et al. 1980).

   The physiological response during diving reflex can be measured by recording standard physiological measures such as heart rate, blood pressure or skin conductance. Heart rate and its interpretation in terms of heart rate variability is becoming more frequently utilized to evaluate the balance between sympathetic and parasympathetic nervous system. Most frequently used is the frequency domain approach which allows differentiating specific frequency bands. The low frequency (LF) band groups the variability between 0.05-0.15Hz and is believed to represent the sympathetic cardiac control with slower unmyelinated nerve fibres while the high frequency (HF) band including frequencies between 0.15-0.4Hz reflects the parasympathetic or vagal control with faster myelinated nerve fibres (Berntson et al 1997).
2. Aims of the study

The aim of the study is to evaluate the effect of a simple vagal manoeuvre, that is a cold face gel mask application, on subjective measures of Anxiety, Disgust, Strength of belief in obsession, Strength of urge to carry out the compulsion, Strength of belief in Theory A/B and an increase in Feeling of being supported, Readiness to face the fear during the ERP treatment of OCD by using a single-case series experimental design and to explore the relationship between subjective measures and sympathovagal balance measured by heart rate variability. Our hypothesis is that:

1. ERP with application of cold gel face mask (Condition B) will be associated with faster reduction of visual analogue scales of Anxiety, Disgust, Strength of belief in obsession, Strength of urge to carry out the compulsion, Strength of belief in Theory A/B and an increase in Feeling of being supported, Readiness to face the fear compared to ERP as usual with simply resisting the compulsive behaviour (Condition C).
2. Increase in vagal tonus as documented by heart rate variability measures will correlate with the effect on visual analogue scales of Anxiety, Disgust, Strength of belief in obsession, Strength of urge to carry out the compulsion, Strength of belief in Theory A/B, Feeling of being supported and Readiness to face the fear.

3. Methods

i. Participants: Participants will be recruited from the Anxiety Disorders Residential Unit (ADRU), Bethlem Royal Hospital. All patients admitted to ADRU have the opportunity to consent to be contacted about participating in research studies. Only patients admitted to ADRU for treatment of OCD who provided such initial consent will be approached by Dr Roman Duncko regarding the written informed consent to participate in the present study.

ii. Procedure and Design: On each day of the study, therapy will begin with the Baseline phase (Condition A) and record the psychological (visual analogue scales of Anxiety, Disgust, Belief in obsession, Strength of urge for compulsion, Strength of belief in Theory A/B, Feeling of being supported, Readiness to face the fear) and physiological measures (HR recording) on 3-5 consecutive 5min intervals or until stable baseline measures are achieved. After that, the participant will proceed with the Intervention phase by applying ERP with the use of triggers as identified on their individual hierarchy. Each ERP session will follow the same structure by first obtaining the session baseline at 3 time points, then exposure to trigger and continue with preventing the response while applying the cold face mask for 5 minutes (Condition B) or without using the face mask (Condition C). Psychological and physiological measures will be obtained in 5 minute intervals until return to session baseline. ERP sessions will follow in alternating order for 4 sessions per day (Day 1: ABCBC, Day 2: ACBCB, Day 3: ABCBC). All baseline and exposure measures will be recorded by the investigator who will by accompanying the participant during the procedure. Cold face gel masks will be stored in refrigerator at the ADRU and will be available to the participant as required.

iii. Psychological measures: Visual analogue scales for measurement of severity of Anxiety, Disgust, Strength of belief in obsession, Strength of urge to carry out the compulsion, Strength of belief in theory A/B, Strength of belief in Theory A/B, Feeling of being supported, Readiness to face the fear will be used by the participant at time points as specified above. In addition to this the participant will be assessed for their clinical symptoms (YBOCS, OCI) on weekly basis as part of their standard treatment plan.

On the last day of the study, participants will be asked to complete the Client Satisfaction Questionnaire based on (Larsen et al 1979) to explore the feasibility and acceptability of the cold face gel mask application during ERP.

iv. Physiological measures: Heart rate variability analysis will be performed on data recorded with a Polar RS800CX heart rate monitor using a H2 chest sensor. Polar monitors have been tested against standard clinical ECG equipment and found to be suitable for heart rate variability analysis (Vanderlei et al 2008). In the morning of the study day, the participants will place the Polar heart rate sensor on their chest using the elastic strap. They will be instructed how to use the heart rate monitor watch Polar RS800CX to record the heart rate and press the mark recording button at specific times during each procedure. At the end of each study day, the data will be downloaded from the heart rate monitor watch and 3 time intervals of 2 minutes will be identified: at the beginning of the condition - time 0, at the beginning of the procedure - time 15, at the end of the condition - time 45. Time intervals will be screened for artefacts and used for heart rate variability analysis using standalone analysis software (Niskanen et al 2004). Variables selected for analysis will include heart rate per minute, time domain measures (RMSSD, NN50) and frequency domain measures (nLF at 0.05-0.15Hz, nHF at 0.15-0.04Hz, LF/HF).

v. Data analysis: Data will be initially evaluated by visual inspection for each participant individually. After that, values obtained for a specific time interval and phase will be averaged among all participants and again evaluated by visual inspection. Percentage of non-overlapping data analysis will be performed to detect statistically significant change between the baseline and intervention phase. Pearson's correlation will be used for correlation analyses.

4. Project timetable

The project is planned to run for 6-12 months depending on the rate of recruitment of participants.

5. Expertise in team

Dr David Veale is a consultant psychiatrist in Cognitive Behaviour Therapy at the South London and Maudsley Trust and a Honorary Senior Lecturer at the Institute of Psychiatry, Kings College London. Specialisms include obsessive compulsive disorder.

Dr Roman Duncko, PhD is a ST5 trainee in General Adult Psychiatry at the South London and Maudsley Trust with long-term research interest in anxiety disorders and autonomic nervous system function.

6. Ethical considerations

All ethical considerations are outlined in the Participant Information and Consent Form that will be distributed to participants. All patients admitted to ARDU who fulfil the inclusion criteria will be approached about participating in the study. All participants will require signing an informed consent to participate. All information and data obtained during the study will be kept in strict confidence. Upon recruitment, every participant will be assigned an anonymous code and the lists linking the code with personal identifying information will be kept secure and separate from the data. Only the Principal Investigator and researchers authorized by the PI will have access to the identifying lists. Every participant will undergo the same procedures with slightly variable order. No deception will be used and participants will be informed as to exactly what the study is about. All participants will be informed at the time of providing consent to participate that they can withdraw from the study at any time and that this will not affect the care they will receive.

7. Dissemination and implementation

Results of the study will be used for poster and/or oral presentations at suitable conferences and for preparing a manuscript for submission in a scientific journal. Depending on the outcome of the study further research will be planned to evaluate the effect of cold face gel mask in a study with randomized control trial design.

ELIGIBILITY:
Inclusion Criteria:

* age over 18 years
* signed informed consent
* established diagnosis of OCD

Exclusion Criteria:

* patients who do not understand English sufficiently to complete the questionnaires
* patients who do not have mental capacity to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2014-07; Primary Completion 2016-02 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
Visual analogue scales at baseline | This measure will be assessed with every exposure on each day of the study at baseline - 5 minutes prior to exposure.
  Rates of Anxiety, Disgust, Strength of belief in obsession, Strength of urge to carry out the compulsion, Strength of belief in theory A/B, Strength of belief in Theory A/B, Feeling of being supported, Readiness to face the fear obtained from visual analogue scales.
Visual analogue scales at exposure | This measure will be assessed with every exposure on each day of the study immediately after finishing the exposure
  Rates of Anxiety, Disgust, Strength of belief in obsession, Strength of urge to carry out the compulsion, Strength of belief in theory A/B, Strength of belief in Theory A/B, Feeling of being supported, Readiness to face the fear obtained from visual analogue scales.
Visual analogue scales 5 minutes post exposure | This measure will be assessed with every exposure on each day of the study at 5 minutes after the exposure.
  Rates of Anxiety, Disgust, Strength of belief in obsession, Strength of urge to carry out the compulsion, Strength of belief in theory A/B, Strength of belief in Theory A/B, Feeling of being supported, Readiness to face the fear obtained from visual analogue scales.
Visual analogue scales 10 minutes post exposure | This measure will be assessed with every exposure on each day of the study at 10 minutes after the exposure.
  Rates of Anxiety, Disgust, Strength of belief in obsession, Strength of urge to carry out the compulsion, Strength of belief in theory A/B, Strength of belief in Theory A/B, Feeling of being supported, Readiness to face the fear obtained from visual analogue scales.
Visual analogue scales 15 minutes post exposure | This measure will be assessed with every exposure on each day of the study at 15 minutes after the exposure.
  Rates of Anxiety, Disgust, Strength of belief in obsession, Strength of urge to carry out the compulsion, Strength of belief in theory A/B, Strength of belief in Theory A/B, Feeling of being supported, Readiness to face the fear obtained from visual analogue scales.

SECONDARY OUTCOMES:
Heart rate variability measures | Heart rate variability measures will be analyzed for specific timeintervals at baseline, during exposure and at three time points after the exposure, at 5, 10 and 15 minutes after exposure.
  Heart rate will be recorded during each ERP session. Hear rate and Heart Rate Variability (HRV) measures will be analyzed in 2 minute intervals corresponding with the timepoints of filling in the VAS at baseline, during the exposure and at three time points after the exposure, at 5, 10 and 15 minutes after the exposure. The Heart Rate Variability measures will include heart rate per minute, time domain measures (RMSSD, NN50) and frequency domain measures (nLF at 0.05-0.15Hz, nHF at 0.15-0.04Hz, LF/HF).

OTHER OUTCOMES:
Symptom severity measures | These measures will be assessed within 1 week prior to the beginning of study and within 1 week after the last ERP session.
  YBOCS and OCI questionnaires
Client Satisfaction Questionnaire | This measure will be assessed within 1 week of completing the study.
  Client Satisfaction Questionnaire used to explore the feasibility and acceptability of the cold face gel mask application during ERP

CONTACTS AND LOCATIONS:
Overall Officials: Roman Duncko, PhD MRCPsych, Principal Investigator — South London and Mausdley NHS Trust
Locations (1):
- Anxiety Disorders Residential Unit, Bethlem Royal Hospital, Beckenham, Kent, United Kingdom

REFERENCES:
- [Background] Arnold RW. The human heart rate response profiles to five vagal maneuvers. Yale J Biol Med. 1999 Jul-Aug;72(4):237-44. PMID 10907774
- [Background] Austin MA, Riniolo TC, Porges SW. Borderline personality disorder and emotion regulation: insights from the Polyvagal Theory. Brain Cogn. 2007 Oct;65(1):69-76. doi: 10.1016/j.bandc.2006.05.007. Epub 2007 Jul 30. PMID 17659821
- [Background] Berntson GG, Bigger JT Jr, Eckberg DL, Grossman P, Kaufmann PG, Malik M, Nagaraja HN, Porges SW, Saul JP, Stone PH, van der Molen MW. Heart rate variability: origins, methods, and interpretive caveats. Psychophysiology. 1997 Nov;34(6):623-48. doi: 10.1111/j.1469-8986.1997.tb02140.x. PMID 9401419
- [Background] Blechert J, Michael T, Grossman P, Lajtman M, Wilhelm FH. Autonomic and respiratory characteristics of posttraumatic stress disorder and panic disorder. Psychosom Med. 2007 Dec;69(9):935-43. doi: 10.1097/PSY.0b013e31815a8f6b. Epub 2007 Nov 8. PMID 17991823
- [Background] Broderick J, Grisham JR, Weidemann G. Disgust and fear responding in contamination-based obsessive-compulsive disorder during pictorial exposure. Behav Ther. 2013 Mar;44(1):27-38. doi: 10.1016/j.beth.2012.05.005. Epub 2012 Jun 8. PMID 23312424
- [Background] Buhlmann U, Wilhelm S, Deckersbach T, Rauch SL, Pitman RK, Orr SP. Physiologic responses to loud tones in individuals with obsessive-compulsive disorder. Psychosom Med. 2007 Feb-Mar;69(2):166-72. doi: 10.1097/PSY.0b013e31802f2799. Epub 2007 Feb 8. PMID 17289827
- [Background] Foa EB. Cognitive behavioral therapy of obsessive-compulsive disorder. Dialogues Clin Neurosci. 2010;12(2):199-207. doi: 10.31887/DCNS.2010.12.2/efoa. PMID 20623924
- [Background] Friedman BH, Thayer JF. Anxiety and autonomic flexibility: a cardiovascular approach. Biol Psychol. 1998 Nov;49(3):303-23. doi: 10.1016/s0301-0511(98)00051-9. PMID 9858059
- [Background] Gooden BA. Mechanism of the human diving response. Integr Physiol Behav Sci. 1994 Jan-Mar;29(1):6-16. doi: 10.1007/BF02691277. PMID 8018553
- [Background] Gorman JM, Sloan RP. Heart rate variability in depressive and anxiety disorders. Am Heart J. 2000 Oct;140(4 Suppl):77-83. doi: 10.1067/mhj.2000.109981. PMID 11011352
- [Background] Hoehn-Saric R, McLeod DR, Hipsley P. Is hyperarousal essential to obsessive-compulsive disorder? Diminished physiologic flexibility, but not hyperarousal, characterizes patients with obsessive-compulsive disorder. Arch Gen Psychiatry. 1995 Aug;52(8):688-93. doi: 10.1001/archpsyc.1995.03950200078017. PMID 7632122
- [Background] Kawano A, Tanaka Y, Ishitobi Y, Maruyama Y, Ando T, Inoue A, Okamoto S, Imanaga J, Kanehisa M, Higuma H, Ninomiya T, Tsuru J, Akiyoshi J. Salivary alpha-amylase and cortisol responsiveness following electrical stimulation stress in obsessive-compulsive disorder patients. Psychiatry Res. 2013 Aug 30;209(1):85-90. doi: 10.1016/j.psychres.2012.11.010. Epub 2012 Dec 23. PMID 23266021
- [Background] Kellner M, Wiedemann K, Yassouridis A, Muhtz C. Non-response of cortisol during stressful exposure therapy in patients with obsessive-compulsive disorder--preliminary results. Psychiatry Res. 2012 Sep 30;199(2):111-4. doi: 10.1016/j.psychres.2012.04.029. Epub 2012 May 11. PMID 22578822
- [Background] Khurana RK, Watabiki S, Hebel JR, Toro R, Nelson E. Cold face test in the assessment of trigeminal-brainstem-vagal function in humans. Ann Neurol. 1980 Feb;7(2):144-9. doi: 10.1002/ana.410070209. PMID 7369721
- [Background] Larsen DL, Attkisson CC, Hargreaves WA, Nguyen TD. Assessment of client/patient satisfaction: development of a general scale. Eval Program Plann. 1979;2(3):197-207. doi: 10.1016/0149-7189(79)90094-6. No abstract available. PMID 10245370
- [Background] Miu AC, Heilman RM, Miclea M. Reduced heart rate variability and vagal tone in anxiety: trait versus state, and the effects of autogenic training. Auton Neurosci. 2009 Jan 28;145(1-2):99-103. doi: 10.1016/j.autneu.2008.11.010. Epub 2008 Dec 6. PMID 19059813
- [Background] National Collaborating Centre for Mental Health (UK). Obsessive-Compulsive Disorder: Core Interventions in the Treatment of Obsessive-Compulsive Disorder and Body Dysmorphic Disorder. Leicester (UK): British Psychological Society (UK); 2006. Available from http://www.ncbi.nlm.nih.gov/books/NBK56458/ PMID 21834191
- [Background] Niskanen JP, Tarvainen MP, Ranta-Aho PO, Karjalainen PA. Software for advanced HRV analysis. Comput Methods Programs Biomed. 2004 Oct;76(1):73-81. doi: 10.1016/j.cmpb.2004.03.004. PMID 15313543
- [Background] Olatunji BO, Lohr JM, Sawchuk CN, Tolin DF. Multimodal assessment of disgust in contamination-related obsessive-compulsive disorder. Behav Res Ther. 2007 Feb;45(2):263-76. doi: 10.1016/j.brat.2006.03.004. Epub 2006 May 12. PMID 16697976
- [Background] Olatunji BO, Wolitzky-Taylor KB, Willems J, Lohr JM, Armstrong T. Differential habituation of fear and disgust during repeated exposure to threat-relevant stimuli in contamination-based OCD: an analogue study. J Anxiety Disord. 2009 Jan;23(1):118-23. doi: 10.1016/j.janxdis.2008.04.006. Epub 2008 May 3. PMID 18541403
- [Background] Ottaviani C, Mancini F, Petrocchi N, Medea B, Couyoumdjian A. Autonomic correlates of physical and moral disgust. Int J Psychophysiol. 2013 Jul;89(1):57-62. doi: 10.1016/j.ijpsycho.2013.05.003. Epub 2013 May 15. PMID 23684734
- [Background] Pittig A, Arch JJ, Lam CW, Craske MG. Heart rate and heart rate variability in panic, social anxiety, obsessive-compulsive, and generalized anxiety disorders at baseline and in response to relaxation and hyperventilation. Int J Psychophysiol. 2013 Jan;87(1):19-27. doi: 10.1016/j.ijpsycho.2012.10.012. Epub 2012 Oct 27. PMID 23107994
- [Background] Stemper B, Hilz MJ, Rauhut U, Neundorfer B. Evaluation of cold face test bradycardia by means of spectral analysis. Clin Auton Res. 2002 Apr;12(2):78-83. doi: 10.1007/s102860200024. PMID 12102454
- [Background] Streeter CC, Gerbarg PL, Saper RB, Ciraulo DA, Brown RP. Effects of yoga on the autonomic nervous system, gamma-aminobutyric-acid, and allostasis in epilepsy, depression, and post-traumatic stress disorder. Med Hypotheses. 2012 May;78(5):571-9. doi: 10.1016/j.mehy.2012.01.021. Epub 2012 Feb 24. PMID 22365651
- [Background] Vanderlei LC, Silva RA, Pastre CM, Azevedo FM, Godoy MF. Comparison of the Polar S810i monitor and the ECG for the analysis of heart rate variability in the time and frequency domains. Braz J Med Biol Res. 2008 Oct;41(10):854-9. doi: 10.1590/s0100-879x2008005000039. Epub 2008 Sep 30. PMID 18853042